CLINICAL TRIAL: NCT01251718
Title: Post-marketing Surveillance of Donepezil Hydrochloride- Investigation of the Clinical Safety and Effectiveness in Patients With Alzheimer's Disease
Brief Title: Post-marketing Surveillance of Donepezil Hydrochloride -Investigation of the Clinical Safety and Effectiveness in Patients With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ART06T
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Donepezil hydrochloride; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Donepezil Hydrochloride
  Interventions: Drug: donepezil hydrochloride

INTERVENTIONS:
Drug: donepezil hydrochloride — Initial dose of 3 mg orally once daily. After 1-2 weeks, dosage increased to 5 mg orally once daily. After 4 or more weeks, dosage increased to 10 mg orally once daily for patients with severe dementia of Alzheimer's type. Dose reduced appropriately according to patient's symptoms.

SUMMARY:
To investigate the clinical safety and effectiveness of donepezil hydrochloride administration in patients with mild or moderate Alzheimer's Disease

ELIGIBILITY:
Inclusion criteria;

Patients diagnosed as Alzheimer's Disease by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).

Patients diagnosed as mild or moderate Alzheimer's Disease, applicable to Functional Assessment Staging (FAST) score 4 or 5.

Exclusion criteria;

Patients who used Aricept within 3 months prior to dosing.

Patients registered this survey before.

Patients with a history of hypersensitivity to any ingredients of Aricept or piperidine derivatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's Disease
Sampling Method: Non-Probability Sample
Enrollment: 894 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2016-02-18 (Actual)

PRIMARY OUTCOMES:
ADAS-Jcog (test of cognitive function) | 36 month (12 weeks and every 6 months)

SECONDARY OUTCOMES:
Adverse events/adverse drug reactions | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Shoya Yamakawa, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (106):
- Japan (106):
  - Anjo, Aichi-ken
  - Nagoya, Aichi-ken
  - Daisen, Akita
  - Hirosaki, Aomori
  - Towada, Aomori
  - Ichihara, Chiba
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Iyo, Ehime
  - Matsuyama, Ehime
  - Niihama, Ehime
  - Tōon, Ehime
  - Kitakyushu, Fukuoka
  - Omuta, Fukuoka
  - Ukiha, Fukuoka
  - Iwaki, Fukushima
  - Mizunami, Gifu
  - Fujioka, Gunma
  - Fukuyama, Hiroshima
  - Kure, Hiroshima
  - Miyoshi, Hiroshima
  - Ōtake, Hiroshima
  - Hakodate, Hokkaido
  - Nayoro, Hokkaido
  - Obihiro, Hokkaido
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Sunagawa, Hokkaido
  - Aioi, Hyōgo
  - Akashi, Hyōgo
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Moriya, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Kita, Kagawa-ken
  - Mitoyo, Kagawa-ken
  - Ebina, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Nankoku, Kochi
  - Uji, Kyoto
  - Suzuka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Sendai, Miyagi
  - Kitamorokata, Miyazaki
  - Iida, Nagano
  - Matsumoto, Nagano
  - Okaya, Nagano
  - Sasebo, Nagasaki
  - Ikoma, Nara
  - Kashihara, Nara
  - Saiki, Oita Prefecture
  - Yufu, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Izumisano, Osaka
  - Kaizuka, Osaka
  - Matsubara, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Fukaya, Saitama
  - Hannō, Saitama
  - Iruma, Saitama
  - Koshigaya, Saitama
  - Sayama, Saitama
  - Masuda, Shimane
  - Hamamatsu, Shizuoka
  - Adachi City, Tokyo
  - Bunkyo, Tokyo
  - Hachiōji, Tokyo
  - Katsushika-ku, Tokyo
  - Machida, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo
  - Nakano City, Tokyo
  - Setagaya City, Tokyo
  - Shinjuku, Tokyo
  - tabashi City, Tokyo
  - Taitō City, Tokyo
  - Toshima City, Tokyo
  - Kurayoshi, Tottori
  - Nanto, Toyama
  - Kinokawa, Wakayama
  - Tendō, Yamagata
  - Hagi, Yamaguchi
  - Shūnan, Yamaguchi
  - Ube, Yamaguchi
  - Akita
  - Chiba
  - Fukuoka
  - Fukushima
  - Gifu
  - Hiroshima
  - Kagoshima
  - Kochi
  - Kyoto
  - Nara
  - Niigata
  - Okayama
  - Osaka
  - Ōita
  - Shizuoka
  - Yamanashi